CLINICAL TRIAL: NCT05583578
Title: Development of a Home-based Self-delivered Prehabilitation Intervention to Proactively Reduce Fall Risk in Older Adults
Brief Title: HOMEStudy: Development of a Home-based Self-delivered Prehabilitation Intervention to Proactively Reduce Fall Risk in Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB202201802; P30AG028740 (NIH)
Record Dates: First submitted 2022-10-13; First posted 2022-10-17 (Actual); Results first posted 2025-01-13 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Mobility Limitation; Aging
MeSH Terms: conditions — Mobility Limitation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Active tDCS (Experimental): Twenty minutes of 2.0mA direct current through two biocarbon rubber electrodes encased in saline soaked 5cm2 sponges placed over the frontal cortices at F3 and F4 (based on the international "10-20 system" of standardized brain electrode placement).
  Interventions: Device: Home-based mobility testing and active tDCS
- Sham tDCS (Sham Comparator): 30 seconds (at the beginning and end of 20 minutes) of 2.0mA direct current through two biocarbon rubber electrodes encased in saline soaked 5cm2 sponges placed over the frontal cortices at F3 and F4 (based on the international "10-20 system" of standardized brain electrode placement).
  Interventions: Device: Sham tDCS

INTERVENTIONS:
Device: Home-based mobility testing and active tDCS — A Soterix Clinical Trials tDCS unit will be used for delivery of stimulation for twenty minutes of 2.0mA direct current through two biocarbon rubber electrodes encased in saline soaked 5cm2 sponges placed over the frontal cortices at F3 and F4 (based on the international "10-20 system" of standardized brain electrode placement). 2.0mA was
  Arms: Active tDCS
Device: Sham tDCS — Sham stimulation is performed with the same device and all procedures will be identical except for the duration of stimulation. Participants will receive 30 seconds of 2.0mA of direct current stimulation at the beginning of each rehabilitation session. Since participants habituate to the sensation of tDCS within 30-60 seconds of stimulation, this procedure provides the same sensation of active tDCS.
  Arms: Sham tDCS

SUMMARY:
Older adults often have difficulty performing complex walking tasks leading to increased fall incidence and subsequent injury. Even in the best clinical settings, it may not be possible for patients or clinicians to dedicate the time and financial resources needed to enact lasting improvements. The study will investigate the use of non-invasive brain stimulation and motor imagery practice within participants homes to assess study design feasibility and potential for mobility improvement.

ELIGIBILITY:
Inclusion Criteria:

* Age 70 - 95 years of age
* Self-report having a risk of falling. Fall risk will be determined by asking whether the participant has had (and recovered from) a fall related injury in the previous year or had fallen two or more times in the previous year or if the participant is afraid of falling because of their balance or walking. (This criterion is based on the 2020 NEJM study: "A Randomized Trial of a Multifactorial Strategy to Prevent Serious Fall Injuries")
* Self-report of "some difficulty with walking tasks, such as becoming tired when walking a quarter mile, or when climbing two flights of stairs, or when performing household chores."
* Willingness to be randomized to either study group and to participate in all aspects of the study assessment and intervention.
* Living in the community and able to travel to the research site.
* Ability to independently assemble and put on the tDCS headband or incorporate the involvement of a willing study partner (e.g., a spouse, family member, or friend) who agrees to assist with this task during each home intervention session.
* Access to an internet-connected computer or television capable of playing videos with sound located in a quiet area with a comfortable stationary chair.
* Able to provide informed consent.

Exclusion Criteria:

* Diagnosed neurological disorder or injury of the central nervous system, or observation of symptoms consistent with such a condition (spinal cord injury, Alzheimer's, Parkinson's, stroke, etc.)
* A score of 23 or lower on the Montreal Cognitive Assessment (MoCA)
* Contraindications to non-invasive brain stimulation (e.g., metal in head, wound on scalp)
* Use of medications affecting the central nervous system including, but not limited to, benzodiazepines, anti-cholinergic medications, and GABAergic medications.
* Severe arthritis, such as awaiting joint replacement
* Current cardiovascular, lung or renal disease; diabetes; terminal illness
* Myocardial infarction or major heart surgery in the previous year
* Cancer treatment in the past year, except for nonmelanoma skin cancers and cancers having an excellent prognosis (e.g., early-stage breast or prostate cancer)
* Current diagnosis of schizophrenia, other psychotic disorders, or bipolar disorder
* Difficulty communicating with study personnel (including people who cannot speak English)
* Uncontrolled hypertension at rest (systolic > 180 mmHg and/or diastolic > 100 mmHg)
* Bone fracture or joint replacement in the previous six months
* Current participation in physical therapy for lower extremity function or cardiopulmonary rehabilitation
* Current enrollment in any clinical trial
* Clinical judgment of investigative team

Ages: 70 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 34 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-02-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clayton Swanson, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Swanson CW, Vial SE, Manini TM, Sibille KT, Clark DJ. Protocol for a home-based self-delivered prehabilitation intervention to proactively reduce fall risk in older adults: a pilot randomized controlled trial of transcranial direct current stimulation and motor imagery. Pilot Feasibility Stud. 2024 Jun 14;10(1):89. doi: 10.1186/s40814-024-01516-1. PMID 38877595

RESULTS

PARTICIPANT FLOW:
Groups:
- Active tDCS: A Soterix mini Clinical Trials tDCS unit will be used for delivery of active stimulation. Participants received twenty minutes of 2.0mA direct current through two biocarbon rubber electrodes encased in saline soaked 5cm2 sponges placed over the frontal cortices at F3 and F4 (based on the international "10-20 system" of standardized brain electrode placement).
- Sham tDCS: A Soterix mini Clinical Trials tDCS unit was used for delivery of sham stimulation. Participants received 30 seconds of 2.0mA of direct current stimulation at the beginning of each 20 minute session. Since participants habituate to the sensation of tDCS within 30-60 seconds of stimulation, this procedure provides the same sensation of active tDCS while only receiving 30 seconds of stimulation at the beginning and end.
Period: Overall Study
Arm/Group | Active tDCS | Sham tDCS
Started | 17 | 17
Completed | 15 | 17
Not Completed | 2 | 0
Not completed — Withdrawal by Subject | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active tDCS | Sham tDCS | Total
Number analyzed (Participants) | 17 | 17 | 34
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 17 | 17 | 34
Age, Continuous [Mean (Standard Deviation); unit: years] | 77.7 (4.06) | 81.0 (5.04) | 79.35 (4.80)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 9 | 17
  Male | 9 | 8 | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 17 | 17 | 34
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 17 | 16 | 33
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 17 | 17 | 34
Height [Mean (Standard Deviation); unit: meters] | 1.69 (0.12) | 1.68 (0.11) | 1.69 (0.11)
Mass [Mean (Standard Deviation); unit: kilograms] | 80.26 (14.01) | 74.21 (16.53) | 77.23 (15.40)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: weight (kg) / [height (m)]2] | 27.9 (3.70) | 26.1 (4.82) | 27.01 (4.33)
Montreal Cognitive Assessment (MoCA) [Mean (Standard Deviation); unit: units on a scale] — Name: Montreal Cognitive Assessment
  Abbreviation: MoCA
  Construct: The MoCA measures global cognitive function.
  Scale Range: 0 to 30
  Interpretation: Higher scores indicate better cognitive function, while lower scores suggest greater cognitive impairment. A score of 26 or higher is typically considered normal, while lower scores may indicate mild cognitive impairment or more severe deficits.
  units on a scale | 26.7 (1.65) | 26.4 (1.80) | 26.53 (1.71)
Activities-specific Balance Confidence (ABC) Scale [Mean (Standard Deviation); unit: units on a scale] — Name: Activities-specific Balance Confidence Scale
  Abbreviation: ABC Scale
  Construct: Assesses an individual's confidence in performing various ambulatory activities without losing balance or becoming unsteady.
  Scale Range: 0% to 100% (each item is rated 0-100, and an average percentage score is calculated)
  Interpretation: Higher scores indicate greater balance confidence, while lower scores suggest lower balance confidence and possible fear of falling.
  units on a scale | 86.6 (9.75) | 86.3 (12.59) | 86.46 (11.09)
Motor Imagery Questionnaire (MIQ-RS) [Mean (Standard Deviation); unit: units on a scale] — Name: Motor Imagery Questionnaire - Revised Second Version
  Abbreviation: MIQ-RS
  Construct: Assesses the ease with which individuals can perform motor imagery tasks in both visual and kinesthetic modalities.
  Scale Range: 7-point Likert scale from 1 = very hard to see/feel to 7 = very easy to see/feel
  Interpretation: Higher scores indicate better ability to engage in motor imagery, while lower scores indicate difficulty in performing mental imagery tasks.
  units on a scale | 6.3 (0.89) | 6.1 (0.75) | 6.21 (0.82)
Katz Index of Independence [Mean (Standard Deviation); unit: units on a scale] — Name: Katz Index of Independence in Activities of Daily Living
  Abbreviation: Katz Index
  Construct: Measures an individual's independence in performing basic activities of daily living (ADLs), such as bathing, dressing, toileting, transferring, continence, and feeding.
  Scale Range: 0 to 6 (1 point per independent activity)
  Interpretation: Higher scores indicate greater independence, while lower scores suggest higher dependence in performing ADLs.
  units on a scale | 6.0 (0) | 5.9 (0.33) | 5.94 (0.24)
Movement-Specific Reinvestment Scale [Mean (Standard Deviation); unit: units on a scale] — Name: Movement-Specific Reinvestment Scale
  Abbreviation: MSRS
  Construct: Assesses the extent to which an individual consciously monitors and controls their movements, potentially disrupting automaticity of movement.
  Scale Range: 10 to 50 (each item is rated on a 5-point Likert scale from 1 = strongly disagree to 5 = strongly agree)
  Interpretation: Higher scores indicate a higher tendency for conscious movement control, which may be associated with poorer movement performance, particularly under pressure.
  units on a scale | 32.6 (10.95) | 33.2 (11.28) | 32.9 (11.0)
Pittsburgh Sleep Quality Index (PSQI) [Mean (Standard Deviation); unit: units on a scale] — Name: Pittsburgh Sleep Quality Index
  Abbreviation: PSQI
  Construct: Assesses sleep quality and disturbances over a 1-month period across several domains, including sleep duration, latency, efficiency, disturbances, medication use, and daytime dysfunction.
  Scale Range: 0 to 21 (global score based on 7 components, each scored 0-3)
  Interpretation: Higher scores indicate worse sleep quality, with a global score greater than 5 suggesting significant sleep disturbances or poor sleep quality.
  units on a scale | 5.3 (2.02) | 6.2 (2.96) | 5.74 (2.54)
Short Form-36 (SF-36): General Health Subscale [Mean (Standard Deviation); unit: units on a scale] — Name: Short Form-36 Health Survey Abbreviation: SF-36 Subscale: General Health Construct: Assesses perceptions of overall health, including personal health status and expectations of future health.
  Subscale Range: 0 to 100 (calculated by transforming raw scores) Interpretation: Higher scores indicate better perceived general health, while lower scores indicate poorer perceived general health.
  Scoring Information: The General Health subscale is calculated by via five items related to overall health perception. The SF-36 does not compute an overall score but eight individual subscales.
  units on a scale | 76.2 (13.29) | 75 (13.11) | 75.6 (13.01)

OUTCOME MEASURES:

1. Primary Outcome: Walking Speed Change From Baseline
Description: Change in the fastest safe walking speed during a two minute walk test
Time Frame: Measured at follow up visit (approximately three weeks after baseline)
Measure: Mean (Standard Error); unit: m/s
Arm/Group | Active tDCS | Sham tDCS
Number analyzed (Participants) | 15 | 17
m/s | 0.052 (0.098) | -0.026 (0.052)
Statistical Analysis 1: Comparison: Active tDCS vs Sham tDCS; Test type: Superiority; p = 0.012, t-test, 2 sided — The Threshold for statistical significance was p=0.05
Statistical Analysis 2: Comparison: Active tDCS vs Sham tDCS; Post-intervention changes in walking speed; Test type: Other; Cohen's d (effect size) = 0.98 — Effect sizes greater than (d = 0.80) were considered large

2. Secondary Outcome: Timed up and go Completion Time From Baseline
Description: Change in the time to complete a 7 meter timed up and go
Time Frame: Measured at follow up visit (approximately three weeks after baseline)
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Active tDCS | Sham tDCS
Number analyzed (Participants) | 15 | 17
seconds | -0.22 (1.70) | 0.31 (1.73)
Statistical Analysis 1: Comparison: Active tDCS vs Sham tDCS; Test type: Superiority; p = 0.39, t-test, 2 sided — The threshold for statistical significance was p = 0.05
Statistical Analysis 2: Comparison: Active tDCS vs Sham tDCS; Test type: Superiority; Cohen's d (effect size) = 0.31 — Effect sizes ranging from 0.21 to 0.79 were considered moderate, anything ≥0.80 were considered large

ADVERSE EVENTS:
Time Frame: The duration in which participants were enrolled in the study to when they completed all study procedures (3 months)
Arm/Group | Active tDCS | Sham tDCS
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/17
Other Adverse Events (participants affected / at risk) | 0/17 | 0/17

LIMITATIONS AND CAVEATS:
This pilot study was primarily designed to evaluate the feasibility and acceptability of a home-based, self-delivered motor imagery intervention for older adults at risk of falling. Consequently, the primary outcomes-changes in walking speed and time to complete the Timed Up and Go (TUG) test-were not intended for inferential statistical analysis. Instead, they were analyzed to provide variance estimates and effect sizes to guide the design of a future follow-up investigation.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-10-18): https://cdn.clinicaltrials.gov/large-docs/78/NCT05583578/Prot_SAP_001.pdf
  • Informed Consent Form (2023-10-18): https://cdn.clinicaltrials.gov/large-docs/78/NCT05583578/ICF_000.pdf